CLINICAL TRIAL: NCT00393211
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, 12-Week Trial to Assess the Efficacy and Safety of MK0663 in Patients With Chronic Low Back Pain
Brief Title: Effect of Etoricoxib to Treat Chronic Low Back Pain (0663-042)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-042; 2006_547
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Etoricoxib; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, Etoricoxib / Duration of Treatment : 12 Weeks
Drug: Comparator : placebo (unspecified) /Duration of Treatment : 12 Weeks

SUMMARY:
Study the effect of etoricoxib 60 mg and 90 mg compared to placebo to treat chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for previous 3 months and majority of days in last month
* Regular use of acetaminophen or NSAID to treat low back pain in past month
* Judged to be in otherwise good health

Exclusion Criteria:

* Low back pain that is due to secondary causes
* Radicular/myelopathic pain
* Surgery for low back pain within the past 6 months
* Active lawsuit or claim pertaining to their low back pain
* Disease that may confound the results of the study or pose risk to the patients
* Corticosteroid use in past month
* Previous participation in an MK0663 study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2000-04; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Low back pain intensity scale (0-100 mm VAS) over 4 weeks compared to placebo

SECONDARY OUTCOMES:
Low back pain intensity scale (0-100 mm VAS) over 12 weeks compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Birbara CA, Puopolo AD, Munoz DR, Sheldon EA, Mangione A, Bohidar NR, Geba GP; Etoricoxib Protocol 042 Study Group. Treatment of chronic low back pain with etoricoxib, a new cyclo-oxygenase-2 selective inhibitor: improvement in pain and disability--a randomized, placebo-controlled, 3-month trial. J Pain. 2003 Aug;4(6):307-15. doi: 10.1016/s1526-5900(03)00633-3. PMID 14622687
- [Background] Curtis SP, Ng J, Yu Q, Shingo S, Bergman G, McCormick CL, Reicin AS. Renal effects of etoricoxib and comparator nonsteroidal anti-inflammatory drugs in controlled clinical trials. Clin Ther. 2004 Jan;26(1):70-83. doi: 10.1016/s0149-2918(04)90007-0. PMID 14996519
- [Background] Sheldon EA, Bird SR, Smugar SS, Tershakovec AM. Correlation of measures of pain, function, and overall response: results pooled from two identical studies of etoricoxib in chronic low back pain. Spine (Phila Pa 1976). 2008 Mar 1;33(5):533-8. doi: 10.1097/BRS.0b013e3181657d24. PMID 18317199